CLINICAL TRIAL: NCT02712554
Title: A Randomized, Double-Blind, Placebo and Active-Controlled, Crossover Study in Opioid-Experienced, Non-Dependent Recreational Drug Users to Determine the Abuse Potential and Safety of CL-108 Tablets Administered Via the Oral Route
Brief Title: A Study in Opioid-Experienced, Non-Dependent Recreational Drug Users to Determine the Abuse Potential and Safety of CL-108 Tablets Administered Via the Oral Route
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Charleston Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CLCT-007
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Pain; Nausea; Vomiting
Keywords: Pain; Nausea; Vomiting
MeSH Terms: conditions — Pain; Nausea; Vomiting | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Treatment A:CL-108 22.5mg/975mg/37.5mg (Experimental): CL-108 22.5 mg/975 mg/37.5 mg tablet by mouth
  Interventions: Drug: CL-108
- Treatment B:CL-108 37.5mg/1625mg/62.5mg (Experimental): CL-108 37.5 mg/1625 mg/62.5 mg tablet by mouth
  Interventions: Drug: CL-108
- Treatment C:M366 22.5mg/975mg (Active Comparator): M366 22.5 mg/975 mg tablet by mouth
  Interventions: Drug: M366
- Treatment D: M366 37.5mg/1625mg (Active Comparator): M366 37.5 mg/1625 mg tablet by mouth
  Interventions: Drug: M366
- Treatment E: Placebo (Placebo Comparator): Placebo 0 mg tablet by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CL-108 — 7.5 mg/325 mg/12.5 mg tablet
  Other Names: Low-dose CL-108 and High-dose CL-108
  Arms: Treatment A:CL-108 22.5mg/975mg/37.5mg; Treatment B:CL-108 37.5mg/1625mg/62.5mg
Drug: M366 — 7.5 mg/325 mg tablet
  Other Names: Low-dose M366 and High-dose M366
  Arms: Treatment C:M366 22.5mg/975mg; Treatment D: M366 37.5mg/1625mg
Drug: Placebo
  Other Names: 0 mg tablet
  Arms: Treatment E: Placebo

SUMMARY:
The purpose of this study is to assess the abuse potential of CL-108 tablets, including the abuse deterrent effects of promethazine, following oral administration, relative to hydrocodone/acetaminophen (APAP) tablets and placebo in non-dependent, recreational opioid users.

DETAILED DESCRIPTION:
The purpose of this study is to assess the abuse potential of CL-108 tablets, including the abuse deterrent effects of promethazine, following oral administration, relative to hydrocodone/acetaminophen (APAP) tablets and placebo in non-dependent, recreational opioid users; to assess the cognitive and behavioral effects of CL-108 tablets following oral administration relative to hydrocodone/APAP tablets and placebo in non-dependent, recreational opioid users; and to assess the safety of orally administered CL-108 tablets relative to hydrocodone/APAP tablets and placebo in non-dependent, recreational opioid users.

ELIGIBILITY:
Inclusion Criteria:

* BMI within 18.0 to 33.0 kg/m2, inclusive (minimum weight of 50.0 kg at Screening)
* Healthy, as determined by no clinically significant medical history, physical examination findings, 12-lead ECG findings, vital signs measurements, and laboratory results at screening, as judged by the investigator
* Current opioid users who had used oral opioids for recreational (non-therapeutic) purposes, at least 10 times in the past year

Exclusion Criteria:

* Drug or alcohol dependence within the last 12 months (except nicotine)
* Subjects who had ever been in treatment for substance use disorders (except smoking cessation
* History of presence of any clinically significant cardiac, neurologic, pulmonary, psychiatric, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, dermatologic, renal, or other major disease at screening, which in the opinion of the investigator, would have jeopardized the safety of the subject or the validity of the study results
* History or presence of hypotension, judged to be clinically significant based on investigator judgement

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard P Schachtel, M.D, Study Chair — Charleston Laboratories

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 12 subjects were enrolled and completed the Dose Selection phase. Subjects randomized to the Treatment phase were 40 and all of them received at least 1 dose of study drug, and 37 subjects completed the study.
Groups:
- Part A (Dose Selection Phase): CL-108 or Placebo: Treatment AA: CL-108 15 mg/650 mg/25 mg tablet by mouth
  Treatment BB: CL-108 22.5 mg/975 mg/37.5 mg tablet by mouth
  Treatment CC: CL-108 30 mg/1300 mg/50 mg tablet by mouth
  Treatment DD: CL-108 37.5 mg/1625 mg/62.5 mg tablet by mouth
  Treatment EE: Placebo 0 mg tablet by mouth
- Part B (Treatment Phase): CL-108, M366 and Placebo: Treatment A (low-dose): CL-108 22.5 mg/975 mg/37.5 mg tablet by mouth
  Treatment B (high-dose): CL-108 37.5 mg/1625 mg/62.5 mg tablet by mouth
  Treatment C (low-dose): M366 22.5 mg/975 mg tablet by mouth
  Treatment D (high-dose): M366 37.5 mg/1625 mg tablet by mouth
  Treatment E: Placebo 0 mg tablet by mouth
Period: Part A: Dose Selection Phase
Arm/Group | Part A (Dose Selection Phase): CL-108 or Placebo | Part B (Treatment Phase): CL-108, M366 and Placebo
Started | 12 | 0
Completed | 12 | 0 (Subjects who participated in Dose Selection Phase were not eligible to participate in Part B.)
Not Completed | 0 | 0
Period: Part B: Qualification Phase
Arm/Group | Part A (Dose Selection Phase): CL-108 or Placebo | Part B (Treatment Phase): CL-108, M366 and Placebo
Started | 0 | 61
Completed | 0 | 40
Not Completed | 0 | 21
Not completed — Drug Discrimination Failure | 0 | 13
Not completed — Sponsor Decision | 0 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 0 | 1
Period: Part B: Treatment Phase
Arm/Group | Part A (Dose Selection Phase): CL-108 or Placebo | Part B (Treatment Phase): CL-108, M366 and Placebo
Started | 0 | 40
Completed | 0 | 37
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (Dose Selection Phase): CL-108 or Placebo | Part B (Treatment Phase): CL-108, M366 and Placebo | Total
Number analyzed (Participants) | 12 | 40 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 40 | 52
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 8 | 32 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 34 | 44
  Black or African American | 1 | 3 | 4
  American Indian or Alaska Native | 0 | 1 | 1
  Multiple | 0 | 2 | 2
  Asian | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 9 | 36 | 45
Region of Enrollment [Number; unit: participants]
  United States | 12 | 40 | 52

OUTCOME MEASURES:

1. Primary Outcome: Subjective Effects: Maximum Effect (Emax) and Minimum Effect (Emin) of High Visual Analog Scale (VAS) in Dose Selection Phase
Description: High VAS measures the positive effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so'). For VAS assessment, pre-dose (baseline) value was subtracted from each post-dose value prior to calculation of the pharmacodynamic (PD) parameter. Emax is the largest effect score and Emin is the smallest effect score between 0 to 24 hours post-dose.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours (post-dose)
Population: Safety population.
  Parameters were not calculated for subjects who experienced emesis within the first 3 hours post-dose.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment AA: CL-108 15 mg/650 mg/25 mg: CL-108 15 mg/650 mg/25 mg tablet by mouth
- Treatment BB: CL-108 22.5 mg/975 mg/37.5 mg: CL-108 22.5 mg/975 mg/37.5 mg tablet by mouth
- Treatment CC: CL-108 30 mg/1300 mg/50 mg: CL-108 30 mg/1300 mg/50 mg tablet by mouth
- Treatment DD: CL-108 37.5 mg/1625 mg/62.5 mg: CL-108 37.5 mg/1625 mg/62.5 mg tablet by mouth
- Treatment EE: Placebo: Placebo 0 mg tablet by mouth
Arm/Group | Treatment AA: CL-108 15 mg/650 mg/25 mg | Treatment BB: CL-108 22.5 mg/975 mg/37.5 mg | Treatment CC: CL-108 30 mg/1300 mg/50 mg | Treatment DD: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment EE: Placebo
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 4
units on a scale
  Emax | 85.0 (21.21) | 42.0 (21.21) | 75.5 (34.65) | 94.0 | 2.3 (4.50)
  Emin | 3.0 (4.24) | 23.5 (3.54) | 42.0 (11.31) | 7.0 | 60.8 (20.84)

2. Primary Outcome: Subjective Effects: Emax of Any Effects VAS in Dose Selection Phase
Description: Any drug effects VAS measures other subjective effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so'). Emax is the largest effect score between 0 (pre-dose) to 24 hours post-dose.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours (post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment AA: CL-108 15 mg/650 mg/25 mg | Treatment BB: CL-108 22.5 mg/975 mg/37.5 mg | Treatment CC: CL-108 30 mg/1300 mg/50 mg | Treatment DD: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment EE: Placebo
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 4
units on a scale | 86.0 (19.80) | 48.5 (26.16) | 75.0 (35.36) | 94.0 | 4.3 (5.68)

3. Primary Outcome: Emax of Drug Liking VAS in Treatment Phase
Description: Drug liking VAS is the measure of balance of effects that assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar (VAS) anchored in the center with a neutral anchor of 'neither like nor dislike' (score of 50 mm), on the left with 'strong disliking' (score of 0 mm) and on the right with 'strong liking' (score of 100 mm). Emax is the largest effect score between 0.5 to 24 hours post-dose.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8 and 24 hours
Population: Intended to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment A: CL-108 22.5 mg/975 mg/37.5 mg: CL-108 22.5 mg/975 mg/37.5 mg tablet by mouth
- Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg: CL-108 37.5 mg/1625 mg/62.5 mg tablet by mouth
- Treatment C: M366 22.5 mg/975 mg: M366 22.5 mg/975 mg tablet by mouth
- Treatment D: M366 37.5 mg/1625 mg: M366 37.5 mg/1625 mg tablet by mouth
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 77.3 (14.68) | 81.4 (13.10) | 74.4 (13.75) | 79.8 (13.07) | 54.5 (9.95)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Test type: Superiority or Other; p = 0.2344, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Test type: Superiority or Other; p = 0.4737, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

4. Secondary Outcome: Number of Adverse Events in Dose Selection Phase
Description: AE=Adverse Event. SAE=Serious adverse event. TEAE=Treatment-emergent adverse event.
Time Frame: Up to visit 3 (Follow up)
Population: Safety population.
Measure: Number; unit: Event
Groups:
- Part A: Dose Selection Phase: Naloxone 0.2 mg bolus intravenously followed by a 10 mL saline flush
  CL-108 15 mg/650 mg/25 mg
  CL-108 22.5 mg/975 mg/37.5 mg
  CL-108 30 mg/1300 mg/50 mg
  CL-108 37.5 mg/1625 mg/62.5 mg
  Placebo 0 mg
Arm/Group | Part A: Dose Selection Phase
Number analyzed (Participants) | 12
Event
  Total number of AEs | 16
  Total Number of TEAEs | 14
  Number of SAEs | 0
  Number of AEs leading to Discontinuation | 0

5. Secondary Outcome: Balance of Effects: Emin of Drug Liking VAS in Treatment Phase
Description: Drug liking VAS is the measure of balance of effects that assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar (VAS) anchored in the center with a neutral anchor of 'neither like nor dislike' (score of 50 mm), on the left with 'strong disliking' (score of 0 mm) and on the right with 'strong liking' (score of 100 mm). Emin is the smallest effect score between 0.5 to 8 hours post-dose.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 49.0 (3.16) | 46.6 (12.16) | 44.8 (11.67) | 46.5 (12.96) | 47.1 (11.42)

6. Secondary Outcome: Balance of Effects: Time-averaged Area Under the Effect Curve (TA_AUE) of Drug Liking VAS in Treatment Phase
Description: TA_AUE is AUE0-8hr divided by time from dosing to the actual time of the 8-hour post-dose assessment using the trapezoidal rule.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 12.071 (10.4456) | 13.772 (10.6773) | 9.773 (12.4254) | 11.162 (12.8093) | 1.183 (5.0571)

7. Secondary Outcome: Balance of Effects: Emax and Emin of Overall Drug Liking VAS in Treatment Phase
Description: Overall drug liking VAS is the measure of balance of effects that assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carryover effects). A 100 mm bipolar VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = 'strong disliking', 50 mm = 'neither like nor dislike', and 100 mm = 'strong liking'). Emax is the largest effect score and Emin is the smallest effect score between 0 to 8 hours post-dose.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale
  Emax | 70.4 (17.77) | 75.8 (17.16) | 65.2 (17.89) | 71.1 (16.81) | 52.2 (8.74)
  Emin | 61.2 (17.07) | 66.7 (19.96) | 57.2 (18.85) | 59.2 (18.50) | 48.7 (9.21)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emax: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emax: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emax: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.1267, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emax: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.1767, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emax: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Emax: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 7: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emin: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p = 0.0119, ANOVA
Statistical Analysis 8: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emin: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p = 0.0025, ANOVA
Statistical Analysis 9: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emin: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.1679, ANOVA
Statistical Analysis 10: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emin: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.0318, ANOVA
Statistical Analysis 11: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emin: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p = 0.0002, ANOVA
Statistical Analysis 12: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Test type: Superiority or Other; p < .0001, ANOVA

8. Secondary Outcome: Balance of Effects: Emax and Emin of Take Drug Again VAS in Treatment Phase
Description: Take drug again VAS is the measure of balance of effects. It is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm bipolar VAS with score ranging from 0 mm to 100 mm (0 mm = 'definitely not', 50 mm = 'do not care', and 100 mm = 'definitely so'). Emax is the largest effect score and Emin is the smallest effect score between 0 to 8 hours post-dose.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale
  Emax | 74.6 (18.98) | 75.2 (18.49) | 68.9 (19.89) | 71.3 (20.51) | 51.1 (12.45)
  Emin | 66.4 (19.85) | 69.3 (21.07) | 60.9 (21.19) | 61.9 (20.68) | 47.5 (12.04)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emax: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emax: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emax: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.0858, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emax: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.2877, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emax: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Emax: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 7: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emin: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p = 0.0009, ANOVA
Statistical Analysis 8: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emin: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p = 0.0001, ANOVA
Statistical Analysis 9: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emin: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.1130, ANOVA
Statistical Analysis 10: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emin: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.0575, ANOVA
Statistical Analysis 11: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emin: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 12: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Emin: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA

9. Secondary Outcome: Positive Effects: Emax of High VAS in Treatment Phase
Description: High VAS measures the positive effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so'). For VAS assessment, pre-dose (baseline) value was subtracted from each post-dose value prior to calculation of the pharmacodynamic (PD) parameter. Emax is the largest effect score between 0 to 8 hours.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (post-dose)
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 58.9 (29.05) | 71.8 (26.07) | 54.6 (28.41) | 67.5 (22.76) | 5.4 (12.92)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emax: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emax: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emax: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.4025, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emax: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.3184, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emax: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Emax: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA

10. Secondary Outcome: Positive Effects: TA_AUE of High VAS in Treatment Phase
Description: as for outcome 6
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (post-dose)
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 1.055 (2.8942) | 27.850 (21.6226) | 36.363 (21.0716) | 24.500 (20.8024) | 32.050 (20.7004)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.2628, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.2262, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA

11. Secondary Outcome: Positive Effects: Emax of Good Effects VAS in Treatment Phase
Description: Good drug effects VAS measures the positive effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so'). Emax is the largest effect score between 0.5 to 8 hours post-dose.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 6.3 (15.06) | 59.3 (29.42) | 68.3 (25.99) | 52.5 (29.35) | 62.2 (23.24)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emax: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emax: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emax: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.1839, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emax: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.1751, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emax: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Emax: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA

12. Secondary Outcome: Positive Effects: TA_AUE of Good Effects VAS in Treatment Phase
Description: as for outcome 6
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 28.108 (22.0759) | 34.894 (20.5885) | 25.541 (23.1053) | 29.327 (19.7001) | 1.140 (2.9074)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.4013, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.0736, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < .0001, ANOVA

13. Secondary Outcome: Negative Effects: Emax of Bad Effects VAS in Treatment Phase
Description: Bad effects VAS measures the negative effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so'). Emax is the largest effect score between 0.5 to 8 hrs.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 14.8 (21.89) | 30.1 (29.35) | 20.1 (20.61) | 36.1 (30.39) | 2.4 (9.68)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emax: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emax: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emax: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.2223, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emax: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.1638, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emax: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p = 0.0041, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Emax: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

14. Secondary Outcome: Negative Effects: TA_AUE of Bad Effects VAS in Treatment Phase
Description: as for outcome 6
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 5.487 (10.5253) | 12.535 (16.0605) | 7.171 (9.8243) | 13.830 (14.9453) | 0.217 (0.9084)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p = 0.0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.2706, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.5507, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p = 0.0047, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

15. Secondary Outcome: Sedative and Other Effects: Emin of Alertness/Drowsiness VAS in Treatment Phase
Description: Alertness/Drowsiness VAS measures the sedative effects. It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of 'neither drowsy nor alert' (score of 50 mm), on the left with 'very drowsy' (score of 0 mm) and on the right with 'very alert' (score of 100 mm). Alertness/Drowsiness VAS was calculated by subtracting pre-dose (baseline) value from each post-dose value. Emin is the smallest effect score between 0 to 8 hours post-dose.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (post-dose)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 25.3 (18.27) | 20.2 (16.44) | 33.3 (17.46) | 27.9 (18.29) | 47.9 (15.69)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emin: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p = 0.0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emin: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emin: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.0014, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emin: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.0080, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emin: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Emin: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

16. Secondary Outcome: Sedative and Other Effects: TA_AUE of Alertness/Drowsiness VAS in Treatment Phase
Description: Alertness/Drowsiness VAS measures the sedative effects. It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of 'neither drowsy nor alert' (score of 50 mm), on the left with 'very drowsy' (score of 0 mm) and on the right with 'very alert' (score of 100 mm). Alertness/Drowsiness VAS was calculated by subtracting pre-dose (baseline) value from each post-dose value. TA_AUE is AUE0-8hr divided by time from dosing to the actual time of the 8-hour post-dose assessment using trapezoidal rule.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (post-dose)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | -12.103 (14.4192) | -16.919 (17.3774) | -6.751 (13.8670) | -8.737 (15.7482) | -0.348 (6.8048)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p = 0.0024, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p = 0.0012, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.0037, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.0011, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

17. Secondary Outcome: Sedative and Other Effects: Emax of Any Effects VAS in Treatment Phase
Description: Any drug effects VAS measures other subjective effects experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (0 mm = 'definitely not') to 'extremely' (100 mm = 'definitely so'). Emax is the largest effect score between 0.5 to 8 hours post-dose.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 62.4 (26.02) | 71.9 (25.85) | 55.4 (27.11) | 68.9 (21.01) | 7.4 (15.98)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; Emax: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Emax: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; Emax: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.0630, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; Emax: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.4436, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; Emax: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; Emax: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

18. Secondary Outcome: Sedative and Other Effects: TA_AUE of Any Effects VAS in Treatment Phase
Description: as for outcome 6
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
units on a scale | 29.720 (21.4816) | 38.504 (20.2062) | 26.371 (20.7356) | 34.030 (19.3426) | 1.537 (3.7125)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.2335, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.1808, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

19. Secondary Outcome: Objective Measures: Change From Baseline in Choice Reaction Time (CRT) in Treatment Phase
Description: CRT is a computerized 5-choice reaction time test in which the subject must press and hold down a touchscreen button at the bottom of the screen. A yellow spot appeared inside one of 5 yellow circles at the top of the screen. Subjects were to respond to the spot as quickly as they could by letting go of the button and touching the circle where the yellow spot appeared. This was repeated for 30 trials. Lower scores indicate better performance.
Time Frame: 0 (Baseline, pre-dose), 1, 2, 4, 8 and 24 hours (post-dose)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
msec
  Baseline (Predose) | 74.0 (103.15) | 51.9 (22.52) | 51.2 (16.83) | 56.8 (28.83) | 55.0 (19.48)
  1 hrs post-dose | -7.0 (104.21) | 9.8 (23.32) | 8.4 (24.48) | 11.1 (46.97) | 3.9 (34.65)
  2 hrs post-dose | 21.7 (160.21) | 45.5 (81.23) | 24.8 (93.63) | 21.2 (55.12) | 8.8 (27.77)
  4 hrs post-dose | 23.4 (155.96) | 38.3 (74.27) | 11.0 (32.97) | 7.9 (27.71) | 5.1 (20.10)
  8 hrs post-dose | -4.6 (104.99) | 29.0 (56.17) | 4.9 (30.03) | 9.0 (45.69) | 4.9 (30.57)
  24 hrs post-dose | -20.6 (103.86) | 4.9 (35.28) | 16.7 (70.86) | 6.3 (46.15) | 4.1 (29.93)

20. Secondary Outcome: Change From Baseline in Number of Errors (Any Errors) in CRT Test in Treatment Phase
Description: CRT is a computerized 5-choice reaction time test in which the subject must press and hold down a touchscreen button at the bottom of the screen. A yellow spot appeared inside one of 5 yellow circles at the top of the screen. Subjects were to respond to the spot as quickly as they could by letting go of the button and touching the circle where the yellow spot appeared. This was repeated for 30 trials. Lower scores indicate better performance. CRT also measures error scores and response accuracy. Any Errors is a combination of incorrect location errors, inaccurate response errors, no response errors, and premature errors.
Time Frame: 0 (Baseline, pre-dose), 1, 2, 4, 8 and 24 hours (post-dose)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Error per msec
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
Error per msec
  Baseline (Predose) | 0.6 (0.86) | 0.4 (0.90) | 0.5 (0.87) | 0.8 (1.09) | 0.90 (0.15)
  1 hrs post-dose | 0.1 (1.29) | 0.1 (1.28) | 0.97 (0.16) | 1.21 (0.20) | 0.70 (0.12)
  2 hrs post-dose | 0.4 (1.48) | 0.9 (1.45) | 0.1 (1.18) | 0.1 (1.33) | 0.2 (0.92)
  4 hrs post-dose | 0.5 (1.30) | 1.4 (2.15) | 0.1 (1.26) | -0.1 (1.36) | 0.1 (1.10)
  8 hrs post-dose | 0.2 (1.95) | 0.9 (2.11) | 0.1 (0.94) | 0.0 (1.21) | 0.1 (0.19)
  24 hrs post-dose | 0.3 (1.49) | -0.1 (0.92) | 0.5 (1.12) | -0.1 (0.91) | 0.1 (1.04)

21. Secondary Outcome: Pupillometry: Maximum Pupil Constriction (MPC)
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. Pupil diameter was measured using electronic pupillometer. Measurements were collected under mesopic lighting conditions. For each subject, every effort was made to use the same eye for all assessments throughout the study. MPC is calculated as smallest observed pupil diameter - baseline pupil diameter.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (post-dose)
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
mm | 2.51 (0.852) | 3.15 (0.783) | 2.34 (0.852) | 2.75 (0.717) | 0.39 (0.537)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; MPC: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; Treatment D: M366 37.5 mg/1625 mg, Treatment E: Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; MPC: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.1268, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; MPC: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p = 0.0014, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; MPC: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; MPC: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

22. Secondary Outcome: Pupillometry: TA_AUE of MPC in Treatment Phase
Description: as for outcome 6
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, and 8 hours (post-dose)
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment A: CL-108 22.5 mg/975 mg/37.5 mg | Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment C: M366 22.5 mg/975 mg | Treatment D: M366 37.5 mg/1625 mg | Treatment E: Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 37 | 37
mm | 1.565 (0.7042) | 2.355 (0.7394) | 1.317 (0.7014) | 1.888 (0.5855) | -0.153 (0.3308)
Statistical Analysis 1: Comparison: Treatment C: M366 22.5 mg/975 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment C (low-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Treatment D: M366 37.5 mg/1625 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment D (high-dose M366) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment C: M366 22.5 mg/975 mg; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Treatment C (low-dose M366); Test type: Superiority or Other; p = 0.0120, ANOVA
Statistical Analysis 4: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment D: M366 37.5 mg/1625 mg; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Treatment D (high-dose M366); Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 5: Comparison: Treatment A: CL-108 22.5 mg/975 mg/37.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment A (low-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: Treatment B: CL-108 37.5 mg/1625 mg/62.5 mg vs Treatment E: Placebo; TA_AUE0-8hr: Treatment B (high-dose CL-108) - Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: Up to visit 3 (Follow up) for Dose Selection phase and Up to Day 24 (Follow up) for Treatment phase
Description: Total 12 subjects in Dose Selection and 40 subjects in Treatment Phase are enrolled and received at least 1 dose of study drug and were included in the Safety population.
Groups:
- Dose Selection AA: CL-108 15 mg/650 mg/25 mg: CL-108 15 mg/650 mg/25 mg tablet by mouth
- Dose Selection BB: CL-108 22.5 mg/975 mg/37.5 mg; Treatment AA: CL-108 22.5 mg/975 mg/37.5 mg: CL-108 22.5 mg/975 mg/37.5 mg tablet by mouth
- Dose Selection CC: CL-108 30 mg/1300 mg/50 mg: CL-108 30 mg/1300 mg/50 mg tablet by mouth
- Dose Selection CC: CL-108 37.5 mg/1625 mg/62.5 mg; Treatment BB: CL-108 37.5 mg/1625 mg/62.5 mg: CL-108 37.5 mg/1625 mg/62.5 mg tablet by mouth
- Dose Selection EE: Placebo; Treatment EE: Placebo: Placebo 0 mg tablet by mouth
- Treatment CC: M366 22.5 mg/975 mg: M366 22.5 mg/975 mg tablet by mouth
- Treatment DD: M366 37.5 mg/1625 mg: M366 37.5 mg/1625 mg tablet by mouth
Arm/Group | Dose Selection AA: CL-108 15 mg/650 mg/25 mg | Dose Selection BB: CL-108 22.5 mg/975 mg/37.5 mg | Dose Selection CC: CL-108 30 mg/1300 mg/50 mg | Dose Selection CC: CL-108 37.5 mg/1625 mg/62.5 mg | Dose Selection EE: Placebo | Treatment AA: CL-108 22.5 mg/975 mg/37.5 mg | Treatment BB: CL-108 37.5 mg/1625 mg/62.5 mg | Treatment CC: M366 22.5 mg/975 mg | Treatment DD: M366 37.5 mg/1625 mg | Treatment EE: Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/4 | 0/40 | 0/39 | 0/38 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/2 | 2/2 | 1/2 | 2/2 | 0/4 | 30/40 | 34/39 | 28/38 | 31/39 | 14/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Selection AA: CL-108 15 mg/650 mg/25 mg (N=2) | Dose Selection BB: CL-108 22.5 mg/975 mg/37.5 mg (N=2) | Dose Selection CC: CL-108 30 mg/1300 mg/50 mg (N=2) | Dose Selection CC: CL-108 37.5 mg/1625 mg/62.5 mg (N=2) | Dose Selection EE: Placebo (N=4) | Treatment AA: CL-108 22.5 mg/975 mg/37.5 mg (N=40) | Treatment BB: CL-108 37.5 mg/1625 mg/62.5 mg (N=39) | Treatment CC: M366 22.5 mg/975 mg (N=38) | Treatment DD: M366 37.5 mg/1625 mg (N=39) | Treatment EE: Placebo (N=39)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 13 | 23 | 14 | 17 | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 4 | 0
Euphoric Mood (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 10 | 13 | 10 | 9 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 3 | 1
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 7 | 11 | 4 | 9 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 6 | 7 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Disturbance in Attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 3 | 5
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 3 | 7 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Feeling Hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 2 | 2 | 1
Feeling of Relaxation (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No